CLINICAL TRIAL: NCT07295431
Title: A Multicenter, Randomized, Double-Blind, Sham-Controlled, Pivotal Clinical Investigation to Evaluate the Efficacy and Safety of the Digital Therapeutic 'BELL-001' for Improving Symptoms in Patients With Insomnia
Brief Title: Sleep Efficacy Randomized Evaluation of a Novel Digital Therapeutic for Insomnia
Acronym: SERENE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BELL Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BELL-001-S-KR-003; BELL-001-S-KR-003 (Other: BELL Therapeutics Inc.)
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Insomnia; Sleep Initiation and Maintenance Disorders
Keywords: Digital Therapeutic; BELL-001; Insomnia Treatment; Auditory stimulation; Biofeedback; Sleep Onset Latency; Sham-Controlled Trial; Autonomic Regulation; Breathing-Synchronized Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, parallel-group, sham-controlled clinical investigation evaluating the efficacy and safety of the digital therapeutic BELL-001 in adults with insomnia.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design. Participants, investigators, care providers, and outcome assessors are blinded to treatment assignment. The sham device is visually identical to the active device but does not deliver the therapeutic algorithm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BELL-001 Digital Therapeutic (Experimental): Participants assigned to the experimental arm will use BELL-001, a smartphone-based digital therapeutic designed to provide personalized auditory stimulation synchronized with the user's breathing pattern. The intervention is administered nightly during the pre-sleep period for 4 weeks. The device delivers an active algorithm intended to reduce pre-sleep hyperarousal and support sleep initiation.
  Interventions: Device: BELL-001 Digital Therapeutic
- Sham Digital Therapeutic (Sham Comparator): Participants assigned to the sham arm will use a visually identical digital device that does not deliver the active therapeutic algorithm. The sham device mimics the user interface and appearance of BELL-001 to maintain blinding but provides non-therapeutic audio output. Participants will use the device nightly during the pre-sleep period for 4 weeks.
  Interventions: Device: Sham Digital Therapeutic

INTERVENTIONS:
Device: BELL-001 Digital Therapeutic — Participants assigned to the experimental arm will use BELL-001, a smartphone-based digital therapeutic designed to provide personalized auditory stimulation synchronized with the user's breathing pattern. Participants will use the device nightly during the pre-sleep period for 4 weeks. The active algorithm delivers respiratory-synchronized auditory feedback intended to reduce pre-sleep hyperarousal and support sleep initiation.
  Arms: BELL-001 Digital Therapeutic
Device: Sham Digital Therapeutic — A sham version of the BELL-001 software that is visually indistinguishable from the active device but lacks the respiratory-synchronized therapeutic algorithm. It provides non-synchronized audio output and serves as the control condition. Used nightly during the pre-sleep period for 4 weeks.
  Arms: Sham Digital Therapeutic

SUMMARY:
This study is a multicenter, randomized, double-blind, sham-controlled clinical investigation designed to evaluate the effectiveness and safety of BELL-001, a digital therapeutic developed to improve symptoms of insomnia. Insomnia is a common sleep disorder that can significantly affect daytime functioning, mood, and overall quality of life. Many patients continue to have difficulties despite lifestyle changes or medication, and safer, non-pharmacological treatment options are increasingly needed.

BELL-001 is a smartphone-based therapeutic that delivers personalized auditory stimulation during the pre-sleep period. The device is intended to promote relaxation and support the transition into sleep by analyzing individual breathing patterns and providing synchronized sound feedback. The study will compare BELL-001 with a sham (placebo-like) digital device that looks identical but does not provide the active therapeutic functions.

Adults diagnosed with insomnia will be randomly assigned to either the BELL-001 group or the sham group. Participants will use the assigned device for four weeks. Throughout the study, sleep-related symptoms, daytime functioning, fatigue, and quality-of-life measures will be assessed. The primary outcome is the change in Insomnia Severity Index (ISI) scores after four weeks of treatment. Safety will be monitored regularly through participant reports and clinical evaluations.

This trial is being conducted at multiple hospitals in Korea and follows ethical guidelines, including review and approval by institutional review boards (IRBs). Participation is voluntary, and all individuals will provide informed consent before any study procedures begin. The results of this study are expected to provide key evidence for the clinical use of a digital, non-pharmacological intervention for adults with insomnia.

DETAILED DESCRIPTION:
Insomnia is a highly prevalent sleep disorder characterized by persistent difficulty with initiating or maintaining sleep, accompanied by daytime impairment such as fatigue, reduced concentration, mood disturbance, and decreased overall functioning. Despite the availability of pharmacologic options and behavioral approaches such as cognitive behavioral therapy for insomnia (CBT-I), many patients experience limited access, inadequate response, concerns about long-term medication dependence, or difficulty adhering to structured behavioral interventions. As a result, there remains a significant clinical need for safe, accessible, non-pharmacological therapies that can effectively address the underlying physiological and psychological factors contributing to insomnia.

BELL-001 is a novel digital therapeutic designed to modulate pre-sleep physiological arousal through personalized auditory stimulation synchronized to an individual's respiratory rhythm. Pre-sleep hyperarousal, including elevated autonomic activation and persistent cognitive or somatic tension, is recognized as a central mechanism in chronic insomnia. BELL-001 analyzes the user's natural breathing pattern through the smartphone microphone and generates real-time auditory feedback aligned with the respiratory phase. This feedback aims to stabilize breathing rhythms, promote parasympathetic activation, reduce sympathetic hyperarousal, and facilitate the transition from wakefulness to sleep. The therapeutic approach is grounded in neurophysiological principles related to interoception, vagal tone modulation, and auditory-respiratory entrainment. Preliminary feasibility and pilot results, including studies conducted at Seoul National University Hospital and Harvard-affiliated centers, suggest that BELL-001 may shorten sleep latency, improve subjective sleep quality, and modulate autonomic markers such as heart rate variability (HRV).

This pivotal, multicenter, randomized, double-blind, sham-controlled clinical investigation has been designed to evaluate the efficacy and safety of BELL-001 for improving insomnia symptoms in adults diagnosed with insomnia disorder. The study is conducted at multiple tertiary hospitals in Korea under Good Clinical Practice (GCP) and institutional review board (IRB) oversight. A total of 114 participants will be enrolled, with competitive enrollment across all sites. Participants who meet eligibility criteria based on clinical diagnosis, screening interviews, and baseline assessments will be randomly assigned in a 1:1 ratio to the active treatment group (BELL-001) or the sham comparator group. The sham device is designed to closely mimic the visual and functional appearance of the active system but does not deliver personalized respiratory-synchronized auditory feedback, ensuring maintenance of blinding for both participants and investigators.

The treatment duration is four weeks. Participants will be instructed to use the assigned intervention during their pre-sleep routine each night. Throughout the study, standardized questionnaires and validated patient-reported outcomes will be administered to assess insomnia severity, daytime sleepiness, fatigue, mood, anxiety, sleep health, and quality of life. These include the Insomnia Severity Index (ISI), Epworth Sleepiness Scale (ESS), Fatigue Severity Scale (FSS), PHQ-9, GAD-7, EQ-5D-5L, sleep diaries, and user satisfaction scales. The primary endpoint is the change in ISI score from baseline to Week 4. Secondary endpoints include changes in daytime functioning, sleep diary metrics, mood and anxiety symptoms, fatigue, quality of life, work productivity, and subjective satisfaction with the intervention. Exploratory endpoints may include analysis of symptom trajectories, subgroup patterns, and predictors of treatment response.

Safety will be continuously evaluated throughout the study by monitoring adverse events, device-related events, and any clinically significant findings during follow-up visits. Given the low-risk nature of the intervention-a non-invasive, non-pharmacological, software-based digital therapeutic-serious safety concerns are not anticipated. Nonetheless, all participating sites will adhere to rigorous reporting standards, and all safety information will be reviewed by the investigators and institutional review boards (IRBs). No independent data monitoring committee is planned due to the low-risk profile of the intervention and the presence of established safety oversight mechanisms.

Randomization and allocation concealment are managed via a centralized system to ensure blinding of participants, investigators, and study staff. All data will be collected in compliance with GCP and stored in validated electronic case report forms (eCRFs). Statistical analyses will be conducted according to a predefined statistical analysis plan, with the primary analysis based on the full analysis set. The trial is powered to detect a clinically meaningful difference in ISI improvement between active and sham groups. Sensitivity analyses and subgroup analyses will further characterize the robustness of the findings.

The overall aim of this pivotal investigation is to generate definitive clinical evidence supporting the regulatory evaluation and potential approval of BELL-001 as a digital therapeutic medical device for the treatment of insomnia in adults. By rigorously evaluating both symptom improvement and safety outcomes in a randomized, sham-controlled design, this study is expected to establish the therapeutic value of a personalized, physiology-based digital intervention. The results have the potential to advance the field of digital therapeutics, expand accessible options for insomnia management, and contribute to a better understanding of how respiratory-synchronized auditory stimulation may modulate pre-sleep arousal and sleep initiation processes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 to 75 years.
* Clinical diagnosis of insomnia disorder according to ICD-11 criteria (non-organic insomnia or sleep initiation/maintenance disorder).
* Insomnia Severity Index (ISI) score ≥ 15 at screening.
* Reports difficulty initiating or maintaining sleep at least 3 nights per week for ≥ 3 months.
* Willing and able to use a smartphone-based digital therapeutic during the pre-sleep period for 4 weeks.
* Able to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Other primary sleep disorders (e.g., obstructive sleep apnea, restless legs syndrome, narcolepsy, circadian rhythm sleep-wake disorders).
* Major psychiatric disorders that may interfere with study assessment (e.g., psychotic disorders, bipolar disorder, severe major depressive episode).
* Substance use disorder, including alcohol or hypnotic misuse, within the past 12 months.
* Use of sleep-inducing medications or CNS-active drugs that cannot be stabilized or discontinued per protocol.
* Significant medical or neurological conditions that may affect sleep or study outcomes (e.g., severe cardiovascular, respiratory, or neurological disease).
* Night-shift workers or individuals with irregular sleep-wake schedules.
* Pregnancy or breastfeeding.
* Participation in another interventional clinical study within the past 30 days.
* Any condition judged by the investigator to interfere with study participation, safety, or data validity.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) Score | Baseline to Week 4
  The primary endpoint is the change in the Insomnia Severity Index (ISI) total score from baseline to Week 4. The ISI is a validated 7-item patient-reported outcome measure assessing nighttime symptoms, sleep satisfaction, and the impact of insomnia on daytime functioning. Higher scores indicate more severe insomnia.

SECONDARY OUTCOMES:
Change in Daytime Sleepiness (Epworth Sleepiness Scale, ESS) | Baseline to Week 4
  Change in ESS score evaluating daytime sleepiness. Higher scores reflect greater sleep propensity.
Change in Fatigue Severity (Fatigue Severity Scale, FSS) | Baseline to Week 4
  Change in FSS score assessing the impact of fatigue on daily functioning.
Change in Depressive Symptoms (PHQ-9) | Baseline to 4 weeks
  Change in PHQ-9 score to evaluate depressive symptom severity.
Change in Anxiety Symptoms (GAD-7) | Baseline to Week 4
  Change in GAD-7 score reflecting the severity of generalized anxiety symptoms.
Change in Health-Related Quality of Life (EQ-5D-5L) | Baseline to 4 weeks
  Change in EQ-5D-5L index score and visual analog scale assessing general health status.
Sleep Diary Outcomes (sSOL, sSQ, sWASO, Number of Awakenings, sSE, sTST) | Baseline to Week 4
  Changes in daily sleep diary parameters recorded during the 4-week treatment period.
  The composite includes:
  Sleep onset latency (sSOL) Subjective sleep quality (sSQ) Wake after sleep onset (sWASO) Number of nocturnal awakenings Sleep efficiency (sSE) Total sleep time (sTST) Sleep diary entries are completed electronically each morning following device use, and weekly averages are compared between baseline and Week 4.
Change in Work Productivity and Activity Impairment (WPAI-GH) | Baseline to Week 4
  Change in absenteeism, presenteeism, and activity impairment related to general health.
User Satisfaction With Device | Week 4
  User-reported satisfaction with usability and perceived benefit of the assigned digital device.

OTHER OUTCOMES:
Responder Rate (≥6-point improvement in ISI) | Baseline to Week 4
  Proportion of participants achieving clinically meaningful ISI reduction

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Young Jung, Principal Investigator — Seoul National University Hospital; Jung-ik Byun, Principal Investigator — Kyung Hee University Hospital at Gangdong; Joon-Sang Sunwoo, Principal Investigator — Kangbuk Samsung Hospital; Kyung-Jin Hwang, Principal Investigator — Kyunghee University Medical Center; Jung-Won Shin, Principal Investigator — CHA Bundang Medical Center; Hye-Yoon Kim, Principal Investigator — Catholic Kwandong University International St. Mary's Hospital
Locations (6):
- South Korea (6):
  - Seoul National University Hospital, Seoul
  - Catholic Kwandong University International St. Mary's Hospital, Seoul
  - CHA Bundang Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Kyung Hee University Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
The sponsor has not yet determined whether individual participant data (IPD) will be shared. Decisions regarding data sharing will consider regulatory requirements, participant privacy protection, and the scientific value of potential data requests. Any future sharing of de-identified data would occur only after appropriate review and in accordance with applicable laws and institutional policies.